CLINICAL TRIAL: NCT04866576
Title: Effect of a Fermented Soy Product on Cognition, Immune Status and Response to Influenza Vaccine in Elderly Men and Women
Brief Title: Effect of a Fermented Soy Product on Cognition, Immune Status and Vaccine
Acronym: IS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Joan Sabate,DrPH, MD, MD, DrPH, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 5210161
Record Dates: First submitted 2021-03-15; First posted 2021-04-30 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Change; Inflammation; Immune Response
Keywords: Fermented Soy; Cognition; Inflammation; Immunity
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: This is a free-living prospective, randomized, double-blind, parallel study design with 31 subjects in free-living conditions. subjects will be randomized to receive either Q CAN powder or placebo powder for 12 weeks.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participants, study personnel and the data analysts will not be aware of which powder is the active powder and which one is the placebo. Only Principle Investigator will be made aware.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Q CAN PLUS POWDER (Experimental): QCAN PLUS POWDER: 2 pouches per day, each pouch contains (12-15 gms of fermented soy powder)
  Interventions: Dietary Supplement: Q CAN PLUS
- Placebo (Placebo Comparator): Sprouted brown rice protein with flavor (provided by BESO Biological Research Inc.)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Q CAN PLUS — Active powder with fermented soy, 2 pouches per day, each pouch contains 12-15 gms of fermented soy
  Arms: Q CAN PLUS POWDER
Dietary Supplement: Placebo — Maltodextrin powder with Whey protein and flavor (provided by BESO Biological Research, Inc.)
  Arms: Placebo

SUMMARY:
The research study will test the effects of Q CAN PLUS powder on the immune, inflammatory and cognitive functions.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of a fermented soy product (Q-CAN), compared to placebo, on the immune, inflammatory and cognitive functions of elderly individuals. The study intervention will be four months in length. sixty two participants , 65 years or older will be randomized to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Elderly men and women, 65 years of age or older
* Ambulatory
* Able to accommodate the intervention food products
* Live in or around Loma Linda to be able to commute to the Nutrition Research Center

Exclusion Criteria:

* Intolerance to soy products
* Immune system insufficiency or disease
* Insulin dependent diabetes mellitus
* Alzheimer's disease
* Dialysis
* Current cancer radiation or chemotherapy
* Prednisone or Prednisolone Therapy greater than 10mg/d

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Changes in immune status measurements | baseline to week 16
  Immune status measurements will be performed using both static and functional tests on whole blood, serum and peripheral blood mononuclear cells (PBMC). Phlebotomy to obtain the needed samples will be performed at baseline (week 0) and at 16 weeks. Changes in immune status include changes in: (a) lymphocyte activity and cytokine production (b) natural killer cells activity, (c) lymphocyte subsets, and (d) inflammatory markers and cytokines.
Changes in lymphocyte activity and cytokine production | baseline to week 16
  Lymphocyte activity and cytokine production will be measured using enzyme-linked immunoassay (ELISA) and flow cytometry. Peripheral blood mononuclear cells (PBMCs) will be incubated and stimulated with or without phytohemagglutinin (PHA) or Lipopolysaccharide (LPS) and the culture supernatant fluids collected and assayed using ELISA for the following cytokines: granulocyte macrophage colony- stimulating Factor (GM-CSF), tumor necrosis factor alpha (TNF-α), interferon gamma (IFN-γ), interleukin 1 beta (IL-1β), interleukin 2 (IL-2), interleukin 6 (IL-6), and interleukin 10 (IL-10).
Changes in lymphocyte subsets | baseline to week 16
  Immunophenotyping will be performed on cryopreserved PBMCs using a flow cytometry. The following markers will be measured: T cytotoxic cells (Tc; CD3+CD8+), T helper cells (Th; CD3+CD4+), B cells (CD19+), NK cells (NK; CD3-CD16+), and regulatory T cells (Treg; CD3+CD4+CD25+Foxp3+).
Changes in inflammatory factors and cytokines | baseline to week 16
  Inflammatory markers in serum will be measured by ELISA and will include C-reactive protein (CRP), E-selectin, Pentraxin 3, Rantes, MCP-1 and Eotaxin.
  Immunophenotyping will be performed on cryopreserved PBMCs using a flow cytometry. The following markers will be measured: T cytotoxic cells (Tc; CD3+CD8+), T helper cells (Th; CD3+CD4+), B cells (CD19+), NK cells (NK; CD3-CD16+), and regulatory T cells (Treg; CD3+CD4+CD25+Foxp3+). Additional characterization of T cells based on naive and memory phenotypes will be determined by corresponding patterns in the expression of CD45RA, CD45RO and CD62L, while different subpopulations of Tregs will be further differentiated by expressions of GITR, CTLA-4 and LAG-3
Changes in complete blood count (CBC) and differential count | baseline to week 16
  CBC and the differential counts will be performed on whole blood with the use of an automated hematology analyzer at a certified clinical facility.
  Immunophenotyping will be performed on cryopreserved PBMCs using a flow cytometry. The following markers will be measured: T cytotoxic cells (Tc; CD3+CD8+), T helper cells (Th; CD3+CD4+), B cells (CD19+), NK cells (NK; CD3-CD16+), and regulatory T cells (Treg; CD3+CD4+CD25+Foxp3+). Additional characterization of T cells based on naive and memory phenotypes will be determined by corresponding patterns in the expression of CD45RA, CD45RO and CD62L, while different subpopulations of Tregs will be further differentiated by expressions of GITR, CTLA-4 and LAG-3

SECONDARY OUTCOMES:
Changes from baseline in global cognitive composite score | baseline to week 16
  The composite score will be calculated using the scores from the tests listed below. We will calculate the standardized scores of each test as the score of each participant minus the group mean and divide by its standard deviation. The composite score is the mean of the standardized scores.
  The 12 tests are: Rey Auditory Verbal Learning Test (RAVLT), Rey-Osterrieth Complex Figure (ROCF), Semantic Fluency (Animals), Boston Naming Test (BNT), Visual Object and Space Perception Battery (VOSP), Block Design section from the Wechsler Adult Intelligence Scale (WAIS-III), Trail Making Test (TMT), FAS Word Fluency, Stroop Color Word Test, Symbol Digit Modalities Test (SMDT) Digit Span from the WAIS-III and Conners Continuous Performance Test (CPT-II).
Changes in the upper respiratory infection questionnaire score | baseline to week 16
  Upper respiratory tract infections will be tracked using the Jackson and Dowling questionnaire as adapted and published by Martineau et al. (2015). The questionnaire will be completed daily by participants, either manually or electronically, throughout the 20-week study period

CONTACTS AND LOCATIONS:
Overall Officials: Joan Sabate, DrPH, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University School of Public Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No